CLINICAL TRIAL: NCT01585922
Title: Noninvasive Positive Pressure Ventilation in Moderate Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Chen Wang, Vice President, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120418BIRM
Record Dates: First submitted 2012-04-20; First posted 2012-04-26 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: noninvasive positive pressure ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

ARMS (2):
- NPPV (Experimental): Use the NPPV to treat moderate ARDS
  Interventions: Procedure: noninvasive positive pressure ventilation (NPPV)
- IMV (Active Comparator): Use invasive mechanical ventilation in treating the patients allocated to this group.
  Interventions: Procedure: invasive mechanical ventilation

INTERVENTIONS:
Procedure: noninvasive positive pressure ventilation (NPPV) — Use NPPV to treat the ARDS patients,and we choose the NPPV ventilators in which the FiO2 can be fixed, for example: the BiPAP Vision or V60 of Phillip Respironics.
  Arms: NPPV
Procedure: invasive mechanical ventilation — Intubate and give invasive mechanical ventilation to the other group patients when they are allocated at once.
  Arms: IMV

SUMMARY:
In order to identify the effect of noninvasive positive pressure ventilation (NPPV) on decreasing inflammatory response, improving the pathophysiological manifestation and reducing the morbidity and mortality in the moderate acute respiratory distress syndrome (ARDS) patients, the investigators conduct this clinical trial comparing NPPV with invasive mechanical ventilation in more than twenty ICUs in China.

ELIGIBILITY:
Inclusion Criteria:

1. acute onset
2. a clinical presentation of respiratory distress
3. arterial oxygen tension/inspired oxygen fraction (PaO2/FiO2) between 200 mmHg to 300 mmHg. The arterial oxygen tension will be measured in fifteen minutes after NPPV (CPAP 5 cmH2O) was used to the patients stably
4. presence of bilateral pulmonary infiltrate on chest radiograph
5. no evidence of left heart failure as assessed by echocardiography and/or a pulmonary artery wedge pressure( PAWP) < 18 mmHg

Exclusion Criteria:

1. age > 70 years or < 18 years
2. PaCO2 > 50mmHg
3. Glasgow Coma Scale (GCS)< 11
4. Upper airway/facial deformity or injury
5. pneumothorax or pneumomediastinum
6. unable to spontaneously clear secretions from their airway
7. respiratory arrest
8. severe ventricular arrhythmia or active myocardial ischemia
9. severe organ dysfunction (including gastrointestinal hemorrhage, disseminated intravascular coagulation, hepatic and renal dysfunction, SOFA score > 1)
10. severe chronic lung diseases(COPD, Asthma or ILD, et al)
11. end-stage patients who are expected to survive less than six months
12. severe abdominal distension
13. refuse to receive NPPV
14. unable to cooperate with NPPV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | From the date of randomization to the date of discharge from ICU and hospital, or to the date of death of all cause, an expected average of 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Beijing Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun B, He H, Wang Z, Qu J, Li X, Ban C, Wan J, Cao B, Tong Z, Wang C. Emergent severe acute respiratory distress syndrome caused by adenovirus type 55 in immunocompetent adults in 2013: a prospective observational study. Crit Care. 2014 Aug 12;18(4):456. doi: 10.1186/s13054-014-0456-6. PMID 25112957